CLINICAL TRIAL: NCT03370458
Title: Lactobacillus Plantarum DR7 for Gut-Brain-Axis Benefits
Acronym: DR7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Clinical Nutrition Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Min-Tze LIONG, Professor Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPeM/17040228
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Placebo and DR7 will be administered via a parallel design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking will be subjected to Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum DR7 (Experimental): Intervention consists of daily administration of 2g probiotic Lactobacillus plantarum DR7, administered daily at a fixed dosage of 9 log CFU/sachet/day and continue for 12 weeks.
  Intervention: Dietary Supplement: Lactobacillus plantarum DR7
  Interventions: Dietary Supplement: Lactobacillus plantarum DR7
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g placebo (no probiotic bacteria), administered daily and continue for 12 weeks.
  Intervention: Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum DR7 — This project aims to study the benefits of probiotics namely Lactobacillus plantarum DR7 for brain health benefits primarily to alleviate stress, among adults in Malaysia aged from 18-60 years. Secondary emphases include respiratory and gastrointestinal health
  Other Names: DR7
  Arms: Lactobacillus plantarum DR7
Dietary Supplement: Placebo — This project aims to study the benefits of probiotics namely Lactobacillus plantarum DR7 for brain health benefits primarily to alleviate stress, among adults in Malaysia aged from 18-60 years. Secondary emphases include respiratory and gastrointestinal health
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Lactobacillus plantarum DR7 for brain health properties, primarily alleviation of stress, among adults in Malaysia aged from 18 to 60 years.

DETAILED DESCRIPTION:
Probiotics are "live microorganisms which, when administered in adequate amounts, can confer health benefits on the host". Probiotics, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases. While numerous microorganisms that may confer health benefits to the host, the most widely studied probiotics are from the Lactobacillus genera. For the past few decades, probiotics have been studied extensively for their beneficial effects mainly on the host's guts. Recently, probiotics are studied for their promising potentials along the gut-brain-axis. The 'gut-brain-axis' is a bidirectional communication system, dynamic for maintaining homeostasis. Many studies show that certain strains of Lactobacillus improved human's health such as reducing the occurrence of diarrhea caused by rotavirus infections, antibiotic treatment, chemotherapy, or lactose intolerance, reduced irritable bowel syndrome symptoms and treating atopic diseases. Lactobacillus have also gained increasing evidences as an effective therapy in preventing respiratory tract infections such as sinusitis, bronchitis and pneumonia. While the precise mechanisms of using Lactobacillus in management of respiratory infections are largely unknown, speculations include: Lactobacillus compete against pathogens; increase the barrier function in respiratory epithelium; immunostimulatory effects by enhancing cellular immunity with increased activity of natural killer cells and macrophages in airways. Lactobacilli, as one of the largest genera for probiotic microorganisms have been researched to alleviate stress, anxiety and/or depression disorders.

Lactobacillus plantarum DR7 was isolated from fresh cow's milk in Penang, Malaysia. In-vitro evaluation has shown that this putative probiotic strain adhere to the criteria of probiotic characteristics; a) resistant towards acid and bile conditions of the upper gastrointestinal tract, b) does not possess antibiotic resistance as per requirement of the European Food Safety Authority (EFSA), c) able to adhere to mucin, d) has antioxidant properties, e) able to utilize prebiotics such as fructooligosaccharide (FOS), inulin and galactooligosaccharide (GOS), e) has a carbon metabolism profile adhering to the general patterns of lactobacilli, and f) possess antimicrobial properties against gastrointestinal pathogens. In-vivo evaluation using rats shown that this putative probiotic strain has gut protection properties; a) modulation of gastrointestinal microbial profile via suppressing gut pathogen populations and increasing the population of lactobacilli, b) decreasing pro-inflammatory cytokines and increasing anti-inflammatory cytokines in the plasma, and c) reducing inflammation in the lower intestines.

All these indicated that Lactobacillus plantarum DR7 has the potential to be an effective probiotic strain that modulate gut health and immunity. In addition, due to the alleviation of gastrointestinal stress, this strain may be beneficial along the gut-brain-axis to promote brain health as well.

Lactobacillus plantarum DR7 and placebo are produced under GMP and HALAL certified manufacturing facility. Probiotic Lactobacillus plantarum DR7 appears as light yellow powder. Sachets are stored away from direct sunlight and in below 30C according to the storage condition recommendations of the manufacturer. Each dose was supplied in an aluminium sachet and all sachets are identical in taste and appearance. Probiotic Lactobacillus plantarum DR7 does not contain any porcine or bovine ingredients.

The product contains Lactobacillus plantarum DR7 and maltodextrin as excipient while placebo contains only maltodextrin.

A total number of 124 healthy adults from age 18 -60 years old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* 18-60 years old
* Willing to commit throughout the experiment
* Have moderate stress and beyond, as per determined by PSS test

Exclusion Criteria:

* Type-1 diabetes (one of the main metabolite of Lactobacillus is acetic acid. Acetic acid has been reported to affect lipid metabolism in the liver and fat digestion in the pancreas in animal studies, and has been applied in obesity studies)
* Long term medication due to certain severe illness (certain medications may interfere with the survivability of Lactobacillus in the gut, for example the interactions between probiotics and warfarin
* HIV/AIDS (there has been no substantial data on the detrimental effects of probiotics on AIDS patients. However, AIDS patient may be immune-compromised in the sense of "leaky gut" that may lead to bacterial translocation, including translocation of Lactobacillus outside the gut environment, into the blood stream)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency (there has been no substantial data on the detrimental effects of probiotics on G6PD deficiency people. However, certain strains of probiotics have been reported to benefit RBC irregularity disorders such as spur cells formation. One of the main mechanisms, involve the alteration of RBC membrane. Although this is a benefit, we are unsure of the effects on G6PD deficiency people, with weaker RBC).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Alleviation of stress | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in alleviation of stress using PSS questionnaire
Alleviation of depression | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in alleviation of depression using DASS42 questionnaire
Enhancement of cognition ability | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in enhancing cognition ability using Cogstate Brief Battery

SECONDARY OUTCOMES:
Alleviation of respiratory tract infections | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in reducing upper respiratory episodes and symptoms using illness symptom chart
Alleviation of gastrointestinal disorders | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in reducing diarrhea incidents using illness symptom chart
Enhancement of immunity | 12 weeks
  To evaluate the potential of oral administration of Lactobacillus plantarum DR7 in enhancing immunity via blood cytokines analyses

CONTACTS AND LOCATIONS:
Overall Officials: MT Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No